CLINICAL TRIAL: NCT04388098
Title: Oral Health Status of Asthmatic Children and Adolescents
Brief Title: Oral Health Status of Asthmatic Children
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, ŞİRİN GÜNER ONUR, Assist. Prof. Dr., Trakya University
Other Study IDs: 2017/210
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Asthma in Children
Keywords: asthma; children; oral health
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthmatic children: Asthmatic children were clinically examined to assess their dental caries experience and periodontal health condition. Stimulated salivary samples were collected and assessed for salivary flow rate, salivary pH and buffering capacity.
  Interventions: Other: Diagnosis of caries experience and periodontal health
- Non-asthmatic children: Non-asthmatic children were clinically examined to assess their dental caries experience and periodontal health condition. Stimulated salivary samples were collected and assessed for salivary flow rate, salivary pH and buffering capacity.
  Interventions: Other: Diagnosis of caries experience and periodontal health

INTERVENTIONS:
Other: Diagnosis of caries experience and periodontal health

SUMMARY:
This study aimed to investigate the dental caries experience, periodontal health and salivary properties of asthmatic and non-asthmatic children ⁄ adolescents.

DETAILED DESCRIPTION:
A total of 108 children aged from 7 to 16 years old were included in this study and equally divided into two groups: Group I (asthmatic children) and Group II (healthy control). All the children were clinically examined to assess their dental caries experience and periodontal health condition. A trained and calibrated examiner (kappa = 0.95) performed the dental caries examination according to World Health Organization (WHO) criteria. Dental caries status was recorded using the number of decayed, missing or filled teeth (dmft/DMFT) and decayed, missing or filled surface (dmfs/DMFS) indices. Periodontal health was assessed by gingival index [GI] and plaque index(PI). An interview was conducted with parents/guardians and a structured questionnaire was employed to parents in addition to medical records. Stimulated salivary samples were collected and assessed for salivary flow rate, salivary pH and buffering capacity.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 7-16
* Asthma diagnosis
* Asthma treatment for at least 1 year
* Under asthma medication
* Healthy controls without any systemic condition

Exclusion Criteria:

* Asthma diagnosis less than a year

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 108 children aged from 7 to 16 years old were included in this study and equally divided into two groups: Group I (asthmatic children) and Group II (healthy control).
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Oral health status | During examination 1 day
  Caries experience of asthmatic and non-asthmatic children was recorded using the number of decayed, missing or filled teeth (dmft/DMFT) and decayed, missing or filled surface (dmfs/DMFS) indices. The gingival index (GI) was used to assess the gingival condition according to the criteria of Loe and Silness as follows: no gingival inflammation (<0.1), mild inflammation (0.1-1.0), moderate inflammation (1.1-1.9), and severe inflammation in case of marked gingival redness and edema with spontaneous bleeding and ulceration (2.0-3.0) Plaque index(PI) was used to assess the amount of dental plaque.The measurement of the state of oral hygiene by Silness-Löe plaque index is based on recording both soft debris and mineralized deposits on the following teeth: A film of plaque adhering to the free gingival margin and adjacent area of the tooth.
salivary flow rate -Salivary characteristics | 5 minutes after saliva collection
  Stimulated salivary samples were collected and assessed for salivary flow rate. Saliva check buffer kit was used for the measurements according to instructions described on the user guide.
salivary pH - Salivary characteristics | 5 minutes after saliva collection
  Stimulated salivary samples were collected and assessed for salivary pH GC saliva check buffer kit was used for the measurements according to instructions described on the user guide.
buffering capacity - Salivary characteristics | 5 minutes after saliva collection
  Stimulated salivary samples were collected and assessed for buffering capacity. GC saliva check buffer kit was used for the measurements according to instructions described on the user guide.